CLINICAL TRIAL: NCT06125015
Title: Unexpected ABR Results in Patients Suspected With Auditory Neuropathy Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Berna Özge MUTLU, Audiologist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-10840098-772.02-3627
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Auditory Neuropathy
MeSH Terms: conditions — Auditory neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hearing Thresholds Assessments — Auditory Neuropathy Spectrum Disorder (ANSD) is a type of hearing disorder that affects the transmission of sound signals from the inner ear to the brain. In individuals with ANSD, the outer hair cells in the cochlea, which are responsible for amplifying sound, typically function properly. However, there is a disruption in the transmission of auditory information from the cochlea to the auditory nerve and then to the brain. It is characterized by a mismatch between the results of objective hearing tests, such as Auditory Brainstem Response (ABR), and subjective hearing experiences. In ABR tests, the responses of the auditory nerve to sounds may be abnormal, while the individual perceives their hearing to be better than suggested by the test results. In this study we showed ANSD patients with abnormal ABR results by using ABR, Otoacoustic Emissions, Tympanometry and behavioral test batteries.

SUMMARY:
This study aimed to assess the clinical evaluations and potential underlying pathologies in patients diagnosed with Auditory Neuropathy Spectrum Disorder (ANSD) who exhibited unusual results in audiological tests. The research involved the retrospective analysis of audiological tests of 11 patients conducted by expert audiologists at Istanbul Medipol Mega Hospital between 2010 and 2020. These patients displayed abnormalities in their Auditory Brainstem Response (ABR) tests. The study sought to investigate patients with ANSD who presented atypical audiological findings, shedding light on the associated clinical aspects and potential causes of such anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Presence of wave V with cochlear microphonics

Exclusion Criteria:

* Type B tympanogram

Ages: 0 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Measuring Hearing Thresholds with Electrophysiological Tests | 6 years
  Participants' hearing thresholds and cochlear microphonics evaluated by using Auditory Brainstem Responses and Otoacoustic Emissions.
Evaluating Middle Ear Pathologies | 6 years
  Participants' middle ear pathologies evaluated by using Tympanometry
Evaluating Hearing Thresholds by Using Behavioral Tests | 6 years
  Participants' reactions to sounds were assessed using Free Field Audiometry or headphones. These evaluations were conducted initially at the time of diagnosis and subsequently after the patients had started using hearing aids.

IPD SHARING:
Plan to Share IPD: No